CLINICAL TRIAL: NCT07333508
Title: 95% Effective Dose (ED95) of Fospropofol Disodium for Adjunctive Sedation During Spinal Anesthesia in Elderly Patients Undergoing Lower Extremity Surgery
Brief Title: Fospropofol Disodium ED95 for Elderly Spinal Anesthesia Sedation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ya-Qun Zhou (Other)
Responsible Party: Sponsor-Investigator, Ya-Qun Zhou, Associate Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LBFED95
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lower Extremity Surgery
Keywords: Fospropofol Disodium; Elderly Patients; Lower Extremity Surgery; Spinal Anesthesia; Adjunctive Sedation; 95% Effective Dose
MeSH Terms: interventions — fospropofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fospropofol Disodium - Sedation ED95 Exploration (Experimental): This arm aims to explore the 95% effective dose (ED95) of fospropofol disodium for sedation in elderly patients undergoing lower extremity surgery with spinal anesthesia.
  Interventions: Drug: Fospropofol Disodium

INTERVENTIONS:
Drug: Fospropofol Disodium — The initial induction dose is 6.0mg/kg, with a dose gradient of 0.5mg/kg (range: 4.0-8.0mg/kg). Sedation success is defined as a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤3 within 3 minutes after drug administration. Dose adjustment follows the k=3 sequential design: ① 3 consecutive successes → next patient receives a 0.5mg/kg lower dose; ② 1 failure → next patient receives a 0.5mg/kg higher dose; ③ 2 consecutive failures → skip the next gradient.
  Immediately after successful induction (MOAA/S ≤3 within 3 minutes), continuous infusion of fospropofol disodium for sedation maintenance will be initiated. The initial maintenance rate is 6.0mg/kg/h, with a gradient of 0.5mg/kg/h (range: 3.0-7.5mg/kg/h). Maintenance success is defined as MOAA/S score ≤3 in ≥4 of 6 assessments (once every 10 minutes). Dose adjustment follows the k=3 sequential design: ① 3 consecutive successes → next patient receives a 0.5mg/kg/h lower rate; ② 1 failure → next patient receives a 0.

SUMMARY:
This study aims to determine the 95% effective dose (ED95) of fospropofol disodium, a new sedative drug, for adjuvant sedation during spinal anesthesia in elderly patients (aged 65 years and older) undergoing lower extremity surgery (e.g., hip/knee replacement, lower limb fracture fixation).

DETAILED DESCRIPTION:
Fospropofol disodium, the only water-soluble propofol prodrug marketed in China, features mild effects on respiratory and circulatory systems, low injection pain, no lipid metabolism-related adverse reactions, and suitable duration of action-making it a promising sedative for elderly patients. However, clinical data on its use in adjuvant sedation during spinal anesthesia are lacking, with no reports on its effective dose in this specific scenario. This prospective sequential trial aims to determine the 95% effective dose (ED95) of fospropofol disodium for sedation induction and maintenance in elderly patients (≥65 years) undergoing lower extremity surgery with spinal anesthesia, providing evidence-based guidance for safe and rational clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years, no gender restriction
* Scheduled for elective lower extremity surgery with spinal anesthesia
* ASA physical status classification Ⅰ-Ⅲ
* BMI 18.5-28.0
* Written informed consent obtained from patients or their guardians

Exclusion Criteria:

* Age <65 years；
* Non-lower extremity surgery or conversion to general anesthesia；
* ASA physical status classification Ⅳ or above；
* BMI <18.5 or >28.0；
* History of drug abuse or alcohol dependence；
* Preoperative use of sedative or analgesic drugs；
* Refusal to participate or inability to sign informed consent；
* Severe arrhythmia or myocardial infarction within 3 months；
* Severe liver or kidney dysfunction；
* Severe respiratory diseases；
* Coagulopathy；
* Uncorrected severe electrolyte disturbance；
* History of mental illness or cognitive impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
95% Effective Dose (ED95) of Fospropofol Disodium for Sedation in Elderly Patients Undergoing Lower Extremity Surgery with Spinal Anesthesia | ① Induction ED95: Assessed at 3 minutes after completion of the fospropofol disodium induction bolus; ② Maintenance ED95: Assessed throughout the intraoperative maintenance phase (6 evaluations, 10 minutes apart).
  The primary outcome is the 95% effective dose (ED95) of fospropofol disodium for adjuvant sedation during spinal anesthesia in elderly patients (≥65 years), including two key components: ① Induction ED95: The intravenous bolus dose at which 95% of patients achieve a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤3 within 3 minutes of administration (dose range: 4.0-8.0mg/kg, gradient: 0.5mg/kg); ② Maintenance ED95: The continuous intravenous infusion rate at which 95% of patients maintain an MOAA/S score ≤3 in ≥4 out of 6 intraoperative assessments (performed every 10 minutes) after successful induction (rate range: 3.0-7.5mg/kg/h, gradient: 0.5mg/kg/h). Both ED95 values (and their 95% confidence intervals [CI]) will be calculated using Probit regression analysis, with sedation success (effective=1, ineffective=0) as the dependent variable and dose/rate as the independent variable.

SECONDARY OUTCOMES:
Induction Onset Time of Fospropofol Disodium | From the start of fospropofol disodium bolus injection to the first achievement of MOAA/S score ≤3, assessed up to 5 minutes.
  The time from the start of fospropofol disodium bolus injection (sedation induction phase) to the first achievement of a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤3.
Recovery Time After Sedation Maintenance Discontinuation | From the moment of maintenance infusion cessation (start of surgical skin closure) to the time when MOAA/S score returns to 5, assessed up to 30 minutes.
  The time from the cessation of fospropofol disodium continuous infusion (start of surgical skin closure) to the recovery of MOAA/S score to 5 (full alertness, rapid response to name called in normal tone).
Incidence of Respiratory Depression | Throughout the sedation period (from induction drug injection to maintenance infusion cessation) and within 10 minutes postoperatively.
  The proportion of patients with respiratory depression, defined as either respiratory rate <8 breaths per minute (bpm) or oxygen saturation (SpO₂) <90% (sustained for ≥10 seconds) during the entire sedation period (induction + maintenance).
Intraoperative Changes in Mean Arterial Pressure (MAP) | Baseline (pre-sedation), 1/3/5 min post-induction, and every 10 minutes during maintenance.
  Change in mean arterial pressure (MAP) relative to baseline value (recorded after lumbar anesthesia stabilization pre-sedation). Key observation points include: 1 minute, 3 minutes, 5 minutes post-induction; and at each MOAA/S assessment time point during maintenance (every 10 minutes). The maximum decrease/increase percentage of MAP from baseline is calculated (e.g., maximum MAP decrease = [(baseline MAP - intraoperative minimum MAP)/baseline MAP] × 100%).
Intraoperative Changes in Heart Rate (HR) | Baseline (pre-sedation), 1/3/5 min post-induction, and every 10 minutes during maintenance.
  Change in heart rate (HR) relative to baseline value (recorded after lumbar anesthesia stabilization pre-sedation). Key observation points include: 1 minute, 3 minutes, 5 minutes post-induction; and at each MOAA/S assessment time point during maintenance (every 10 minutes). The maximum decrease/increase percentage of HR from baseline is calculated (e.g., maximum HR decrease = [(baseline HR - intraoperative minimum HR)/baseline HR] × 100%).
Incidence of Postoperative Adverse Reactions | Within 24 hours postoperatively (assessed during ward rounds or follow-up).
  The proportion of patients experiencing adverse reactions within 24 hours postoperatively, including:
  Cardiovascular reactions: Hypertension (SBP >160 mmHg or increase of ≥30% from baseline), tachycardia (HR >100 bpm); Gastrointestinal reactions: Nausea, vomiting; Neurological/psychological reactions: Postoperative agitation (restlessness, inability to cooperate with nursing care), dizziness; Others: Injection site pain, pruritus, paresthesia (recorded if persistent for ≥24 hours postoperatively).

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Qun Zhou, Principal Investigator — Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China.
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No